CLINICAL TRIAL: NCT00348374
Title: A Phase 3b, Randomized, Open-Label, Parallel Group, Multicenter Trial Assessing The Efficacy Of Exubera Vs. Lispro Introduced Into A Lantus Based Regimen In Suboptimally Controlled Patients With Type 2 Diabetes Mellitus
Brief Title: Exubera vs Lispro in a Lantus-based Regimen for Improved Glycemic Control in Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A2171093
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Results first posted 2010-03-16 (Estimated); Last update posted 2010-03-16 (Estimated); Status verified 2009-07

CONDITIONS: Diabetes Mellitus
Keywords: type two diabetes, insulin, HbA1c
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance | interventions — Insulin Lispro; Exubera

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insulin Lispro (Active Comparator): Weight based initiation dose, and individually adjusted doses, per subject's blood glucose, over the six months study, in addition to insulin glargine and oral agents.
  Interventions: Drug: Insulin Lispro
- Exubera (Experimental): Weight based initiation dose, and individually adjusted doses, per subject's blood glucose, over the six months study, in addition to insulin glargine and oral agents.
  Interventions: Drug: Exubera

INTERVENTIONS:
Drug: Insulin Lispro — Weight based initiation dose, and individually adjusted doses, per subject's blood glucose, over the six months study, in addition to insulin glargine and oral agents.
  Arms: Insulin Lispro
Drug: Exubera — Weight based initiation dose, and individually adjusted doses, per subject's blood glucose, over the six months study, in addition to insulin glargine and oral agents.
  Arms: Exubera

SUMMARY:
The current trial will examine the efficacy and safety of Exubera administered as a mealtime insulin compared to lispro, when added to an existing regimen of basal insulin glargine + or = Oral Agents (OAs). Dose titrations will be provided which should allow a large proportion of subjects to reach target glycosylated hemoglobin (A1C) levels.

ELIGIBILITY:
Inclusion Criteria:

* Adults with type 2 diabetes using Lantus® (insulin glargine) as their basal insulin, not at glycemic goal.

Exclusion Criteria:

* lung disease
* current smoking or discontinued smoking within past 6 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2006-06; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (59):
- United States (58):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Mobile, Alabama
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Malvern, Arkansas
  - Pfizer Investigational Site, Foot Hill Ranch, California
  - Pfizer Investigational Site, Fresno, California
  - Pfizer Investigational Site, Greenbrae, California
  - Pfizer Investigational Site, Los Gatos, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, San Mateo, California
  - Pfizer Investigational Site, Tustin, California
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, New Britain, Connecticut
  - Pfizer Investigational Site, Washington D.C., District of Columbia
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, West Palm Beach, Florida
  - Pfizer Investigational Site, Winter Park, Florida
  - Pfizer Investigational Site, Columbus, Georgia
  - Pfizer Investigational Site, Decatur, Georgia
  - Pfizer Investigational Site, Honolulu, Hawaii
  - Pfizer Investigational Site, Honululu, Hawaii
  - Pfizer Investigational Site, Idaho Falls, Idaho
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Gurnee, Illinois
  - Pfizer Investigational Site, Des Moines, Iowa
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Bethesda, Maryland
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Flint, Michigan
  - Pfizer Investigational Site, Minneapolis, Minnesota
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, East Syracuse, New York
  - Pfizer Investigational Site, Greenville, North Carolina
  - Pfizer Investigational Site, Morehead City, North Carolina
  - Pfizer Investigational Site, Statesville, North Carolina
  - Pfizer Investigational Site, Kettering, Ohio
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Tulsa, Oklahoma
  - Pfizer Investigational Site, Bend, Oregon
  - Pfizer Investigational Site, Bensalem, Pennsylvania
  - Pfizer Investigational Site, Greenville, South Carolina
  - Pfizer Investigational Site, Bartlett, Tennessee
  - Pfizer Investigational Site, Memphis, Tennessee
  - Pfizer Investigational Site, Arlington, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, El Paso, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Bennington, Vermont
  - Pfizer Investigational Site, Norfolk, Virginia
  - Pfizer Investigational Site, Virginia Beach, Virginia
  - Pfizer Investigational Site, Renton, Washington
  - Pfizer Investigational Site, Spokane, Washington
  - Pfizer Investigational Site, Milwaukee, Wisconsin
- Pfizer Investigational Site, San Juan, Puerto Rico

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A2171093&StudyName=Exubera%20vs%20Lispro%20in%20a%20Lantus-based%20Regimen%20for%20improved%20glycemic%20control%20in%20Type%202%20Diabetes

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 62 centers between June 2006 and August 2008.
Groups:
- Exubera®: Weight based initiation dose of Exubera® (total daily dose: body weight in kilograms (kg) x 0.15 milligrams per kilogram (mg/kg); approx. 0.05 mg/kg per meal, three times per day [TID]), and individually titrated doses per subject's blood glucose in addition to insulin glargine and oral agents.
- Insulin Lispro: Weight based initiation dose of insulin-lispro (total daily dose: body weight in kilograms (kg) x 0.15 milligrams per kilogram (mg/kg); divided into 3 equal preprandial doses [before breakfast, lunch, and dinner], and individually titrated doses per subject's blood glucose, in addition to insulin glargine and oral agents. The approximate insulin-lispro dose in units was prescribed based on the calculated dose of Exubera® (conversion from milligrams (mg) of Exubera® to international units (IU) of insulin-lispro was approx. 3:1).
Period: Overall Study
Arm/Group | Exubera® | Insulin Lispro
Started | 88 | 103
Received Study Treatment | 88 | 96
Completed | 69 | 71
Not Completed | 19 | 32
Not completed — Adverse Event | 1 | 4
Not completed — Lost to Follow-up | 1 | 3
Not completed — Withdrawal by Subject | 5 | 5
Not completed — Other | 11 | 12
Not completed — ongoing at date of cutoff | 1 | 1
Not completed — randomized but did not receive treatment | 0 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exubera® | Insulin Lispro | Total
Number analyzed (Participants) | 88 | 96 | 184
Age, Customized [Number; unit: participants]
  18-44 years | 16 | 19 | 35
  45-64 years | 56 | 51 | 107
  >=65 years | 16 | 26 | 42
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 37 | 74
  Male | 51 | 59 | 110

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin A1c (HbA1c) at End of Treatment
Description: Change from Baseline in glycosylated hemoglobin A1c (HbA1c %) at Week 24. Change = mean value at Week 24 minus mean value at Baseline.
Time Frame: Baseline, Week 24 (End of Treatment)
Population: Full analysis set (FAS): subjects who received at least one dose of study medication, had a baseline glycosylated hemoglobin A1c (HbA1c%) measurement, and had a post-baseline HbA1C measurement; last (post-baseline) observation carried forward (LOCF). Number of subjects with HbA1c values at Baseline and Week 24: Exubera® n=81, Lispro n=90.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Exubera® | Insulin Lispro
Number analyzed (Participants) | 81 | 90
percent | -1.4 (1.3) | -1.6 (1.0)

2. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin A1c (HbA1c) at Each Visit
Description: Change in mean glycosylated hemoglobin A1c (HbA1c %) from Baseline to each visit through Week 24. Change = mean value at observation minus mean value at Baseline.
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24
Population: FAS; LOCF; N=number of subjects with evaluable data; n=number of subjects with evaluable data at observation: Exubera, Lispro, respectively.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Exubera® | Insulin Lispro
Number analyzed (Participants) | 81 | 90
percent
  Week 4 (n=74, 87) | -0.8 (0.7) | -0.8 (0.6)
  Week 8 (n=80, 90) | -1.1 (0.9) | -1.2 (0.9)
  Week 12 (n=81, 90) | -1.3 (1.1) | -1.5 (1.0)
  Week 16 (n=81, 90) | -1.4 (1.1) | -1.5 (1.1)
  Week 20 (n=81, 90) | -1.4 (1.2) | -1.6 (1.1)
  Week 24 (n=81, 90) | -1.4 (1.3) | -1.6 (1.0)

3. Secondary Outcome: Subjects That Attained Glycosylated Hemoglobin A1c (HbA1c) < 7.0%, < 6.5% and < 6.0% at Week 24
Description: Number of subjects acheiving glycemic control: HbA1c target levels of <7.0%, <6.5%, and <6.0% at Week 24.
Time Frame: Week 24
Population: FAS; N=number of subjects with evaluable data at Baseline; n=number of subjects with evaluable data at observation: Exubera, Lispro, respectively.
Measure: Number; unit: participants
Arm/Group | Exubera® | Insulin Lispro
Number analyzed (Participants) | 81 | 90
participants
  HbA1c < 6.0% (n=61, 64) | 8 | 9
  HbA1c < 6.5% (n=61, 64) | 24 | 27
  HbA1c < 7.0% (n=61, 64) | 33 | 41

4. Secondary Outcome: Subjects That Attained Glycosylated Hemoglobin A1c (HbA1c) Target Levels of <7%, < 6.5%, and < 6.0% Without an Episode of Severe Hypoglycemia at Week 24
Description: Number of subjects that attained HbA1c target levels of <7%, < 6.5%,and <6.0% at Week 24 without an episode of severe hypoglycemia.
Time Frame: Week 24
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Exubera® | Insulin Lispro
Number analyzed (Participants) | 81 | 90
participants
  HbA1c < 6.0% (n=61, 63) | 8 | 8
  HbA1c <6.5% (n=61, 63) | 24 | 26
  HbA1c <7% (n=61, 63) | 33 | 40

5. Secondary Outcome: Change From Baseline in Fasting and 2-hour Postprandial Glucose as Determined by 8-point Self-monitored Blood Glucose Profiles
Description: Mean change from Baseline in fasting and 2-hour postprandial glucose at each visit in 8-point self-monitored blood glucose (SMBG) profiles: includes values prior to each meal (breakfast, lunch and dinner), 2 hours after each meal, at bedtime, and at 2:00 ante meridiem (a.m.) Change=observation value minus Baseline value.
Time Frame: Week 1, Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24
Population: FAS; N=number of subjects with evaluable data; n=number of subjects with evaluable data at observation: Exubera, Lispro, respectively.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Exubera® | Insulin Lispro
Number analyzed (Participants) | 81 | 90
mg/dL
  Week 1: Pre-Breakfast [fasting] (n=67, 74) | 11.1 (54.1) | 9.3 (54.3)
  Week 1: 2 Hours Post-Breakfast (n=62, 72) | -36.3 (78.9) | -19.3 (77.5)
  Week 1: 2 Hours Post-Lunch (n=62, 73) | -32.2 (76.2) | -27.9 (84.2)
  Week 1: 2 Hours Post-Supper (n=61, 68) | -30.7 (74.6) | -32.5 (89.5)
  Week 2: Pre-Breakfast [fasting] (n=66, 69) | 5.7 (53.5) | 5.5 (58.4)
  Week 2: 2 Hours Post-Breakfast (n=58, 68) | -43.7 (80.7) | -40.8 (99.3)
  Week 2: 2 Hours Post-Lunch (n=59, 69) | -28.1 (73.4) | -52.0 (92.0)
  Week 2: 2 Hours Post-Supper (n=62, 67) | -32.6 (80.0) | -54.3 (84.9)
  Week 4: Pre-Breakfast [fasting] (n=66, 73) | -2.5 (52.6) | -4.3 (61.9)
  Week 4: 2 Hours Post-Breakfast (n=62, 68) | -50.0 (85.0) | -48.5 (87.0)
  Week 4: 2 Hours Post-Lunch (n=60, 74) | -45.8 (80.1) | -52.4 (96.0)
  Week 4: 2 Hours Post-Supper (n=57, 70) | -44.9 (85.3) | -71.5 (99.0)
  Week 8: Pre-Breakfast [fasting] (n=67, 69) | -6.7 (67.0) | -20.8 (48.6)
  Week 8: 2 Hours Post-Breakfast (n=61, 69) | -50.2 (89.8) | -59.0 (78.8)
  Week 8: 2 Hours Post-Lunch (n=60, 69) | -42.9 (78.5) | -61.0 (95.7)
  Week 8: 2 Hours Post-Supper (n=60, 68) | -45.1 (87.8) | -86.5 (98.5)
  Week 12: Pre-Breakfast [fasting] (n=57, 73) | -12.2 (63.3) | -22.2 (63.0)
  Week 12: 2 Hours Post-Breakfast (n=51, 70) | -46.8 (81.1) | -74.8 (84.3)
  Week 12: 2 Hours Post-Lunch (n=49, 71) | -49.1 (87.6) | -60.6 (98.9)
  Week 12: 2 Hours Post-Supper (n=52, 69) | -48.2 (84.3) | -81.6 (81.5)
  Week 16: Pre-Breakfast [fasting] (n=55, 66) | -26.1 (59.9) | -16.9 (62.0)
  Week 16: 2 Hours Post-Breakfast (n=50, 65) | -55.2 (81.3) | -60.5 (81.7)
  Week 16: 2 Hours Post-Lunch (n=50, 65) | -56.0 (74.9) | -69.9 (99.2)
  Week 16: 2 Hours Post-Supper (n=51, 61) | -53.4 (83.3) | -90.6 (96.1)
  Week 20: Pre-Breakfast [fasting] (n=57, 60) | -25.4 (60.7) | -26.3 (59.9)
  Week 20: 2 Hours Post-Breakfast (n=51, 59) | -64.2 (67.3) | -78.5 (70.7)
  Week 20: 2 Hours Post-Lunch (n=51, 60) | -50.7 (71.1) | -74.1 (91.5)
  Week 20: 2 Hours Post-Supper (n=50, 55) | -62.4 (73.4) | -78.7 (83.9)
  Week 24: Pre-Breakfast [fasting] (n=56, 55) | -26.6 (64.7) | -27.6 (43.9)
  Week 24: 2 Hours Post-Breakfast (n=51, 55) | -61.8 (69.5) | -75.1 (66.3)
  Week 24: 2 Hours Post-Lunch (n=50, 56) | -59.6 (69.9) | -65.5 (94.0)
  Week 24: 2 Hours Post-Supper (n=52, 54) | -58.1 (73.2) | -78.0 (82.2)

6. Secondary Outcome: Change From Baseline in Fasting and Postprandial Plasma Glucose as Determined by Standardized Meal Tolerance Tests at Week 12
Description: Change from Baseine in fasting and postprandial plasma glucose as determined by standardized meal tolerance tests (MTT). Change = mean value at Week 12 minus mean value at Baseline. Time 0 results are for MTT (time 0) and non MTT (implied time 0) subjects.
Time Frame: Baseline, Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Exubera® | Insulin Lispro
Number analyzed (Participants) | 81 | 90
mg/dL
  0 mins (Fasting) (n=25, 42) | -49.8 (68.6) | -30.5 (58.2)
  30 mins (n=6, 6) | -27.9 (65.4) | -44.4 (33.3)
  60 mins (n=23, 35) | -58.8 (75.1) | -50.3 (73.2)
  90 mins (n=25, 38) | -62.8 (73.5) | -69.5 (65.7)
  120 mins (n=26, 40) | -56.3 (71.5) | -77.4 (68.3)
  180 mins (n=26, 37) | -49.1 (79.1) | -76.4 (68.8)

7. Secondary Outcome: Change From Baseline in Fasting and Postprandial Plasma Glucose as Determined by Standardized Meal Tolerance Tests at Week 24
Description: Change from Baseline in fasting and postprandial plasma glucose as determined by standardized meal tolerance tests (MTT). Change = mean value at Week 24 minus mean value at Baseline. Time 0 results are for MTT (time 0) and non MTT (implied time 0) subjects.
Time Frame: Baseline, Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Exubera® | Insulin Lispro
Number analyzed (Participants) | 81 | 90
mg/dL
  0 mins (Fasting) (n=22, 30) | -25.1 (109.5) | -34.8 (64.3)
  30 mins (n=1, 7) | -59.5 (0.0) | -86.0 (43.5)
  60 mins (n=21, 26) | -64.9 (107.9) | -59.8 (61.9)
  90 mins (n=22, 28) | -72.1 (98.9) | -73.6 (54.0)
  120 mins (n=23, 29) | -74.2 (95.0) | -75.7 (59.7)
  180 mins (n=21, 28) | -64.1 (95.9) | -74.2 (66.2)

8. Secondary Outcome: Change From Baseline in Fasting and Postprandial Lipids as Determined by Standard Meal Tolerance Tests
Description: Change from Baseline in fasting and postprandial lipids at Week 12 and Week 24 as determined by standard meal tolerance tests. Change = value at observation minus value at Baseline. Postprandial = 120 mins after meal.
Time Frame: Baseline, Week 12, Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Exubera® | Insulin Lispro
Number analyzed (Participants) | 81 | 90
mg/dL
  Total cholesterol: Week 12 Fasting (n=60, 79) | -4.4 (21.1) | 1.2 (34.9)
  Total cholesterol: Week 12 Postprandial(n=22, 33) | -6.8 (14.8) | -6.7 (31.2)
  Total cholesterol: Week 24 Fasting (n=51, 59) | -0.2 (31.7) | 0.5 (29.9)
  Total cholesterol Week 24 Postprandial(n=17, 21) | 0.7 (34.3) | -4.7 (29.5)
  HDL cholesterol: Week 12 Fasting (n=60, 79) | 1.2 (4.5) | 1.4 (5.5)
  HDL cholesterol: Week 12 Postprandial (n=22, 33) | 1.3 (3.5) | 1.1 (5.3)
  HDL cholesterol: Week 24 Fasting (n=51, 59) | 1.1 (5.2) | 0.4 (5.9)
  HDL cholesterol: Week 12 Postprandial (n=17, 21) | 0.0 (5.7) | -0.4 (6.0)
  LDL cholesterol: Week 12 Fasting (n=60, 79) | 1.3 (19.8) | 5.9 (29.3)
  LDL cholesterol: Week 12 Postprandial (n=22, 33) | -1.4 (13.3) | -1.5 (26.8)
  LDL cholesterol: Week 24 Fasting (n=51, 59) | 3.5 (27.0) | 5.0 (23.9)
  LDL cholesterol: Week 24 Postprandial (n=17, 21) | 2.5 (31.3) | -0.7 (19.9)
  Triglycerides: Week 12: Fasting (n=60, 79) | -34.7 (59.3) | -30.7 (74.3)
  Triglycerides: Week 12 : Postprandial (n=22, 33) | -34.1 (42.8) | -31.6 (71.4)
  Triglycerides: Week 24: Fasting (n=51, 59) | -24.3 (59.3) | -24.9 (98.4)
  Triglycerides: Week 24: Postprandial (n=17, 21) | -9.5 (45.9) | -17.9 (89.0)

9. Secondary Outcome: Number of Subjects With Change From Baseline in Fasting and Postprandial Markers of Cardiovascular (CV) Risk as Determined by Standardized Meal Tolerance Tests
Description: Cardiovascular risk markers included serum high-sensitivity C-reactive protein (hs-CRP)[mg/L], leptin (ng/mL), adiponectin (ug/mL), and spot urine microalbumin. Change = observation of mean fasting and postprandial markers of cardiovascular risk at Week 12 and Week 24 minus mean Baseline observation.
Time Frame: Week 12, Week 24
Population: Due to cancellation of the EXUBERA program, too few patients participated to explore the markers of cardiovascular (CV) risks so these markers were not summarized.
Measure: Number; unit: participants
Arm/Group | Exubera® | Insulin Lispro
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Change From Baseline Weight at Each Visit
Description: Change = mean body weight at observation minus mean body weight at Baseline.
Time Frame: Baseline, Week 1, Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24
Population: FAS; LOCF (all visits except Baseline); N=number of subjects with evaluable data; n=number of subjects with evaluable data at observation: Exubera, Lispro, respectively.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Exubera® | Insulin Lispro
Number analyzed (Participants) | 81 | 90
kilograms
  Week 1 Body weight (n=76, 87) | -0.5 (8.4) | -0.3 (5.9)
  Week 2 Body weight (n=80, 90) | 0.5 (1.5) | 0.9 (1.7)
  Week 4 Body weight (n=81, 90) | 0.1 (8.5) | 0.9 (6.2)
  Week 8 Body weight (n=81, 90) | 1.3 (3.4) | 2.1 (3.1)
  Week 12 Body weight (n=81, 90) | 0.6 (9.9) | 2.3 (3.5)
  Week 16 Body weight (n=81, 90) | 2.5 (3.0) | 2.8 (3.9)
  Week 20 Body weight (n=81, 90) | 2.4 (3.1) | 2.9 (7.0)
  Week 24 Body weight (n=81, 90) | 1.4 (8.4) | 3.8 (4.3)

11. Secondary Outcome: Change From Baseline in Fasting Plasma Lipids
Description: Change from baseline in fasting plasma lipids at Week 12 and Week 24. Change = observation mean minus Baseline mean.
Time Frame: Baseline, Week 12, Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Exubera® | Insulin Lispro
Number analyzed (Participants) | 81 | 90
mg/dL
  Total cholesterol: Week 12 (n=60, 79) | -4.4 (21.1) | 1.2 (34.9)
  Total cholesterol: Week 24 (n=51, 59) | -0.2 (31.7) | 0.5 (29.9)
  HDL cholesterol: Week 12 (n=60, 79) | 1.2 (4.5) | 1.4 (5.5)
  HDL cholesterol: Week 24 (n=51, 59) | 1.1 (5.2) | 0.4 (5.9)
  LDL cholesterol: Week 12 (n=60, 79) | 1.3 (19.8) | 5.9 (29.3)
  LDL cholesterol: Week 24 (n=51, 59) | 3.5 (27.0) | 5.0 (23.9)
  Triglycerides: Week 12 (n=60, 79) | -34.7 (59.3) | -30.7 (74.3)
  Triglycerides: Week 24 (n=51, 59) | -24.3 (59.3) | -24.9 (98.4)

12. Secondary Outcome: Change From Baseline in Insulin Glargine Dose at Each Visit (Office and/or Phone)
Description: Change from Baseline in insulin glargine at each visit. Change = mean at observation minus mean Baseline observation. Basal dose = injection of basal insulin (IU) (insulin glargine).
Time Frame: Baseline, Week 1, Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24
Population: Safety population: all subjects who received at least one dose of study medication; Lispro international units (IU) were converted to milligrams (mg) equivalent; N=number of subjects with evaluable data; n=number of subjects with evaluable data at observation: Exubera, Lispro, respectively.
Measure: Mean (Standard Deviation); unit: IU
Arm/Group | Exubera® | Insulin Lispro
Number analyzed (Participants) | 88 | 96
IU
  Week 1 (n=69, 77) | 8.8 (22.7) | 4.3 (8.9)
  Week 2 (n=60, 69) | 14.1 (24.9) | 9.1 (14.0)
  Week 4 (n=65, 79) | 12.8 (21.2) | 14.0 (11.7)
  Week 8 (n=65, 73) | 16.1 (25.6) | 19.2 (15.6)
  Week 12 (n=57, 68) | 24.9 (26.2) | 21.3 (20.7)
  Week 16 (n=48, 60) | 28.1 (30.7) | 24.3 (21.4)
  Week 20 (n=50, 50) | 31.2 (27.4) | 28.5 (31.6)
  Week 24 (n=29, 38) | 37.1 (33.2) | 31.2 (28.1)

13. Secondary Outcome: Baseline Prandial Insulin Dose (at Each Meal) at Each Visit
Description: Dose of inhaled insulin prior to each meal at each visit.
Time Frame: Week 0, Week 1, Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24
Population: Safety population: all subjects who received at least one dose of study medication; N=number of subjects with evaluable data; n=number of subjects with evaluable data at observation.
Measure: Mean (Standard Deviation); unit: mg
Groups:
- Exubera®: Weight based initiation dose, and individually adjusted doses, per subject's blood glucose, over the six months study, in addition to insulin glargine and oral agents.
Arm/Group | Exubera®
Number analyzed (Participants) | 88
mg
  Week 0: Pre-breakfast (n=81) | 4.14 (1.39)
  Week 0: Pre-lunch (n=86) | 4.10 (1.37)
  Week 0: Pre-dinner (n=87) | 4.06 (1.33)
  Week 1: Pre-breakfast (n=87) | 4.25 (1.45)
  Week 1: Pre-lunch (n=87) | 4.33 (1.42)
  Week 1: Pre-dinner (n=87) | 4.35 (1.49)
  Week 2: Pre-breakfast (n=87) | 4.89 (1.63)
  Week 2: Pre-lunch (n=87) | 4.94 (1.72)
  Week 2: Pre-dinner (n=87) | 5.09 (1.82)
  Week 4: Pre-breakfast (n=84) | 5.44 (2.16)
  Week 4: Pre-lunch (n=84) | 5.46 (2.32)
  Week 4: Pre-dinner (n=84) | 5.71 (2.36)
  Week 8: Pre-breakfast (n=80) | 6.09 (2.93)
  Week 8: Pre-lunch (n=80) | 6.11 (2.99)
  Week 8: Pre-dinner (n=80) | 6.41 (3.07)
  Week 12: Pre-breakfast (n=74) | 6.40 (3.17)
  Week 12: Pre-lunch (n=74) | 6.51 (3.35)
  Week 12: Pre-dinner (n=74) | 7.01 (3.67)
  Week 16: Pre-breakfast (n=71) | 6.69 (3.60)
  Week 16: Pre-lunch (n=71) | 6.78 (3.82)
  Week 16: Pre-dinner (n=71) | 7.40 (4.04)
  Week 20: Pre-breakfast (n=68) | 7.01 (4.06)
  Week 20: Pre-lunch (n=68) | 7.10 (4.20)
  Week 20: Pre-dinner (n=68) | 7.58 (4.30)
  Week 24: Pre-breakfast (n=66) | 7.53 (4.78)
  Week 24: Pre-lunch (n=66) | 7.70 (4.69)
  Week 24: Pre-dinner (n=66) | 7.83 (4.81)

14. Secondary Outcome: Number of Subjects With Hypoglycemic Events
Description: Severe event = subject unable to treat self, at least 1 neurological symptom (memory loss, confusion, uncontrollable/irrational behavior, difficulty awakening, suspected seizure, loss of consciousness), and blood glucose <= 49 milligrams per deciliter (mg/dL) or not measured but clinical manifestations reversed by oral carbohydrates or glucose. Non-severe events = events that were mild-moderate.
Time Frame: Month 1, Month 2, Month 3, Month 4, Month 5, Month 6
Population: Safety population: all subjects who received at least one dose of study medication; N=number of subjects with evaluable data; n=number of subjects with evaluable data at observation: Exubera, Lispro, respectively.
Measure: Number; unit: participants
Arm/Group | Exubera® | Insulin Lispro
Number analyzed (Participants) | 88 | 96
participants
  Month 1: Overall (n=88, 96) | 38 | 35
  Month 1: Mild/Moderate (n=88, 96) | 38 | 35
  Month 1: Severe (n=88, 96) | 0 | 0
  Month 2: Overall (n=81, 91) | 26 | 29
  Month 2: Mild/Moderate (n=81, 91) | 25 | 29
  Month 2: Severe (n=81, 91) | 1 | 0
  Month 3: Overall (n=74, 87) | 29 | 38
  Month 3: Mild/Moderate (n=74, 87) | 29 | 38
  Month 3: Severe (n=74, 87) | 0 | 0
  Month 4: Overall (n=71, 81) | 22 | 28
  Month 4: Mild/Moderate (n=71, 81) | 22 | 28
  Month 4: Severe (n=71, 81) | 0 | 0
  Month 5: Overall (n=69, 75) | 25 | 26
  Month 5: Mild/Moderate (n=69, 75) | 25 | 26
  Month 5: Severe (n=69, 75) | 0 | 0
  Month 6: Overall (n=66, 70) | 17 | 21
  Month 6: Mild/Moderate (n=66, 70) | 17 | 21
  Month 6: Severe (n=66, 70) | 0 | 1

15. Secondary Outcome: Number of Total Hypoglycemic Events
Description: Total number and severity of hypoglycemic events. Severe events = subject unable to treat self, at least 1 neurological symptom (memory loss, confusion, uncontrollable or irrational behavior, difficulty awakening, suspected seizure, loss of consciousness), and blood glucose <= 49 milligrams per deciliter (mg/dL) or not measured but clinical manifestations reversed by oral carbohydrates or glucose. Non-severe events = events that were mild or moderate.
Time Frame: Month 1, Month 2, Month 3, Month 4, Month 5, Month 6
Population: as for outcome 14
Measure: Number; unit: events
Arm/Group | Exubera® | Insulin Lispro
Number analyzed (Participants) | 88 | 96
events
  Month 1: Overall (n=88, 96) | 106 | 121
  Month 1: Mild/Moderate (n=88, 96) | 106 | 121
  Month 1: Severe (n=88, 96) | 0 | 0
  Month 2: Overall (n=81, 91) | 73 | 120
  Month 2: Mild/Moderate (n=81, 91) | 72 | 120
  Month 2: Severe (n=81, 91) | 1 | 0
  Month 3: Overall (n=74, 87) | 103 | 114
  Month 3: Mild/Moderate (n=74, 87) | 101 | 113
  Month 3: Severe (n=74, 87) | 0 | 0
  Month 4: Overall (n=71, 81) | 57 | 80
  Month 4: Mild/Moderate (n=71, 81) | 57 | 80
  Month 4: Severe (n=71, 81) | 0 | 0
  Month 5: Overall (n=69, 75) | 70 | 89
  Month 5: Mild/Moderate (n=69, 75) | 70 | 88
  Month 5: Severe (n=69, 75) | 0 | 0
  Month 6: Overall (n=66, 70) | 35 | 48
  Month 6: Mild/Moderate (n=66, 70) | 35 | 47
  Month 6: Severe (n=66, 70) | 0 | 1

16. Secondary Outcome: Treatment Exposure for Hypoglycemic Subjects at Each Interval of the Study: Number of Subject Months of Treatment
Description: Subject months of treatment = number of days from start of treatment to last day of active treatment + 1 day lag (total number of subjects treated * days treated), including off-drug time)/30.44. Severity: severe = subject unable to treat self, had at least 1 neurological symptom (memory loss, confusion, uncontrollable/irrational behavior, difficulty awakening, suspected seizure, loss of consciousness), and blood glucose <= 49 milligrams/deciliter; or not measured but clinical manifestations were reversed by oral carbohydrates or glucose. Non-severe events = events that were mild or moderate.
Time Frame: Month 1, Month 2, Month 3, Month 4, Month 5, Month 6
Population: as for outcome 14
Measure: Number; unit: subject months of treatment
Arm/Group | Exubera® | Insulin Lispro
Number analyzed (Participants) | 88 | 96
subject months of treatment
  Month 1: Overall (n=88, 96) | 85.3 | 92.9
  Month 1: Mild/Moderate (n=88, 96) | 85.3 | 92.9
  Month 1: Severe (n=88, 96) | 85.3 | 92.9
  Month 2: Overall (n=81, 91) | 78.3 | 88.8
  Month 2: Mild/Moderate (n=81, 91) | 78.3 | 88.8
  Month 2: Severe (n=81, 91) | 78.3 | 88.8
  Month 3: Overall (n=74, 87) | 72.2 | 85.1
  Month 3: Mild/Moderate (n=74, 87) | 72.2 | 85.1
  Month 3: Severe (n=74, 87) | 72.2 | 85.1
  Month 4: Overall (n=71, 81) | 70.4 | 77.6
  Month 4: Mild/Moderate (n=71, 81) | 70.4 | 77.6
  Month 4: Severe (n=71, 81) | 70.4 | 77.6
  Month 5: Overall (n=69, 75) | 68.0 | 73.6
  Month 5: Mild/Moderate (n=69, 75) | 68.0 | 73.6
  Month 5: Severe (n=69, 75) | 68.0 | 73.6
  Month 6: Overall (n=66, 70) | 41.4 | 43.8
  Month 6: Mild/Moderate (n=66, 70) | 41.4 | 43.8
  Month 6: Severe (n=66, 70) | 41.4 | 43.8

17. Secondary Outcome: Crude Hypoglycemic Event Rate
Description: Crude event rate = (number of events)/(subject months); severe hypoglycemic events: crude event rate = (number of events)/(100 subject months). Severe = subject unable to treat self, at least 1 neurological symptom (memory loss, confusion, uncontrollable or irrational behavior, difficulty awakening, suspected seizure, loss of consciousness), and blood glucose <= 49 milligrams per deciliter (mg/dL) or unmeasured but clinical manifestestation reversed by oral carbohydrates or glucose. Non-severe events = mild-moderate.
Time Frame: Month 1, Month 2, Month 3, Month 4, Month 5, Month 6
Population: Safety population; N=number of subjects with evaluable data; n=number of subjects with evaluable data at observation: Exubera, Lispro, respectively.
Measure: Number; unit: events per subject months
Arm/Group | Exubera® | Insulin Lispro
Number analyzed (Participants) | 88 | 96
events per subject months
  Month 1: Overall (n=88, 96) | 1.2 | 1.3
  Month 1: Mild/Moderate (n=88, 96) | 1.2 | 1.3
  Month 1: Severe (n=88, 96) | 0.0 | 0.0
  Month 2: Overall (n=81, 91) | 0.9 | 1.4
  Month 2: Mild/Moderate (n=81, 91) | 0.9 | 1.4
  Month 2: Severe (n=81, 91) | 1.3 | 0.0
  Month 3: Overall (n=74, 87) | 1.4 | 1.3
  Month 3: Mild/Moderate (n=74, 87) | 1.4 | 1.3
  Month 3: Severe (n=74, 87) | 0.0 | 0.0
  Month 4: Overall (n=71, 81) | 0.8 | 1.0
  Month 4: Mild/Moderate (n=71, 81) | 0.8 | 1.0
  Month 4: Severe (n=71, 81) | 0.0 | 0.0
  Month 5: Overall (n=69, 75) | 1.0 | 1.2
  Month 5: Mild/Moderate (n=69, 75) | 1.0 | 1.2
  Month 5: Severe (n=69, 75) | 0.0 | 0.0
  Month 6: Overall (n=66, 70) | 0.8 | 1.1
  Month 6: Mild/Moderate (n=66, 70) | 0.8 | 1.1
  Month 6: Severe (n=66, 70) | 0.0 | 2.3

18. Secondary Outcome: Change From Baseline in Patient Treatment Satisfaction (as Assessed by Patient Satisfaction With Insulin Treatment [PSIT] Questionnaire)
Description: Patient Satisfaction with insulin treatment Questionnaire (PSIT): 15-item self administered questionnaire that measures global satisfaction and two domains (subscales): convenience/ease of use and social comfort in people with type 1 and type 2 diabetes. 5-point Likert scale ranging from 1 (strongly agree) to 5 (strongly disagree). The scoring of responses to each item is analyzed so that a higher item score indicates more satisfaction. Change = mean Patient Satisfaction of Insulin Treatment (PSIT) score at observation minus mean score at Baseline.
Time Frame: Week 4, Week 24
Population: Due to cancellation of the EXUBERA program descriptive statistics for the Patient Satisfaction of Insulin Treatment (PSIT) Questionnaire were not provided.
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | Exubera® | Insulin Lispro
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Change in Patient Treatment Satisfaction (as Assessed by Patient Satisfaction With Insulin Treatment [PSIT] Questionnaire) From Week 4 to Week 24
Description: Patient Satisfaction with insulin treatment Questionnaire (PSIT): 15-item self administered questionnaire that measures global satisfaction and two domains (subscales): convenience/ease of use and social comfort in people with type 1 and type 2 diabetes. 5-point Likert scale ranging from 1 (strongly agree) to 5 (strongly disagree). The scoring of responses to each item is analyzed so that a higher item score indicates more satisfaction.
  Change = difference in mean Patient Satisfaction with Insulin Treatment (PSIT) score from Week 4 to Week 24.
Time Frame: Week 4, Week 24
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | Exubera® | Insulin Lispro
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Change From Baseline in 24-hour Mean Glucose Values Measured by Continuous Glucose Monitoring System (CGMS)
Description: Mean of 24-hour Continuous Glucose Monitoring (CGMS) glucose values. Change from Baseline = mean at observation minus mean Baseline value.
Time Frame: Baseline, Week 12, Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Exubera® | Insulin Lispro
Number analyzed (Participants) | 81 | 90
mg/dL
  Week 12 (n=19, 16) | -30.4 (44.3) | -33.0 (41.9)
  Week 24 (n=17, 13) | -19.4 (43.7) | -23.4 (43.1)

21. Secondary Outcome: Change From Baseline in Standard Deviation of 24-hour Glucose Values Measured by Continuous Glucose Monitoring System (CGMS)
Description: Mean change in standard deviation of all blood glucose values within 24-hour period. Change = mean at observation minus mean at Baseline.
Time Frame: Baseline, Week 12, Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Exubera® | Insulin Lispro
Number analyzed (Participants) | 81 | 90
mg/dL
  Week 12 (n=19, 16) | -3.4 (25.5) | 2.3 (20.9)
  Week 24 (n=17, 13) | -3.6 (22.4) | -0.9 (14.3)

ADVERSE EVENTS:
Description: Number of participants at risk for serious and other adverse events was determined by the number of participants who took at least one dose of study drug.
Arm/Group | Exubera® | Insulin Lispro
Serious Adverse Events (participants affected / at risk) | 3/88 | 3/96
Other Adverse Events (participants affected / at risk) | 68/88 | 67/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exubera® (N=88) | Insulin Lispro (N=96)
Ileus (Gastrointestinal disorders) | 0 | 1
Labyrinthitis (Infections and infestations) | 0 | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Medical device complication (Injury, poisoning and procedural complications) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Exubera® (N=88) | Insulin Lispro (N=96)
Palpitations (Cardiac disorders) | 3 | 5
Vision blurred (Eye disorders) | 4 | 5
Diarrhoea (Gastrointestinal disorders) | 0 | 6
Hunger (General disorders) | 1 | 5
Influenza (Infections and infestations) | 5 | 4
Nasopharyngitis (Infections and infestations) | 5 | 3
Sinusitis (Infections and infestations) | 5 | 3
Upper respiratory tract infection (Infections and infestations) | 9 | 9
Hypoglycaemia (Metabolism and nutrition disorders) | 58 | 59
Dizziness (Nervous system disorders) | 9 | 15
Headache (Nervous system disorders) | 8 | 7
Tremor (Nervous system disorders) | 10 | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 9 | 12

LIMITATIONS AND CAVEATS:
Due to cancellation of the EXUBERA program the sample size was too small to adequately address the inferential objectives of this study. Descriptive statistics for the PSIT Questionnaire and the markers of cardiovascular risk were not provided.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.